CLINICAL TRIAL: NCT01640470
Title: A Multi-Site Trial of the Impact of Assistive Technology With Individuals With Mobility Limitations and Their Caregivers.
Brief Title: A Multi-Site Trial of the Impact of Assistive Technology With Assistance Users and Their Caregivers
Acronym: CATS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal (Other)
Collaborators: Simon Fraser University (Other); Duke University (Other); University of Ottawa (Other)
Responsible Party: Principal Investigator, Louise Demers, Directrice, Département de l'ergothérapie, Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 232262
Record Dates: First submitted 2011-11-21; First posted 2012-07-13 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Mobility Disability; Older Adults; Community Dwelling
Keywords: assistive technology; environmental modification; caregiver; client-centred

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Assistive technology (Experimental): The home based AT Provision, Updating and Tune-Up (ATPUT) Intervention will include recommendations for assistive technology, possibly entailing financial assistance to repair or to acquire new AT, and training. New equipment will likely include devices such as bathroom grab bars, raised toilet seats, walkers, and bath chairs.
  Interventions: Device: Assistive Technology Provision and Tune-Up Intervention
- Customary care (Active Comparator): Participants in this arm will receive customary care.
  Interventions: Device: Customary Care

INTERVENTIONS:
Device: Assistive Technology Provision and Tune-Up Intervention — The home based AT Provision, Updating and Tune-Up (ATPUT) Intervention will consist of 5 components: 1) identification and prioritization of problematic activities by the assistance user and his/her principal, cohabitating caregiver; 2) in-residence assessment of the daily activities and social participation and preferences of the assistance user; 3) detailed review of the AT and human assistance that are currently being used; 4) recommendations by an occupational therapist for possible changes in the personal assistance strategy; 5) negotiation of an ATPUT Personal Plan with the assistance user and her/his principal caregiver.
  The intervention occurs over a six week period and involves 3 to 6 visits from an occupational therapist.
  Arms: Assistive technology
Device: Customary Care — Participants in the customary care group receive normal occupational therapy services.Occupational Therapy
  Other Names: Customary device prescription and training
  Arms: Customary care

SUMMARY:
Many individuals with mobility limitations, especially those who are older and have more severe impairments, use a combination of assistive devices and personal assistance to meet their needs. Assistive technology (AT), which includes devices such as wheelchairs, walkers, bathroom grab bars, and dressing aids, helps facilitate day-to-day activities and social participation (basic and instrumental activities of daily living) among these individuals and may decrease their dependence on human assistance. Although some research has reported beneficial outcomes of AT use, few studies have used controlled experimental designs. Furthermore, the results are often difficult to interpret because the AT interventions are only vaguely described. Another concern is that many individuals receive help from others, but scant attention has been paid to the impact of AT on caregivers. This neglect produces an incomplete portrayal of the effect of AT interventions. The proposed study addresses these deficiencies by evaluating the effects of a formalized dyadic AT intervention on individuals with mobility limitations and on their caregivers. The Assistive Technology Provision, Updating and Training (ATPUT)intervention involves a detailed in-home assessment of participants' current AT; the negotiation and implementation of a personal AT plan with the participants and their caregivers; and the provision of AT devices, non-structural home modifications, and device training.

Objectives:

1. To determine the efficacy of the Assistive Technology Provision, Updating and Training intervention for assistance users and for their caregivers.
2. To explore how the intervention is experienced by these individuals and to help explain the study findings.

General Hypotheses:

The investigators anticipate this intervention will increase the daily activities and social participation of individuals with mobility limitations; decrease the psychological and physical demands on caregivers; and reduce the amount of caregiving required.

Methodologies:

This research will use a combination of quantitative and qualitative methods. The quantitative portion will be an experimental, single-blinded study in which the investigators randomly assign participants to either the ATPUT or a customary care group.

ELIGIBILITY:
Inclusion Criteria:

* daily activity and/or mobility disability
* referred to homecare
* have an unpaid informal caregiver who is above the age of consent and willing to participate in the study
* can communicate in English or French.

Exclusion Criteria:

* cognitive impairments that are likely to prevent them from reliably completing the study questionnaires.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2011-12; Primary Completion 2016-05 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Caregiver Assistive Technology Outcome Measure | 58 Weeks
  The caregiver assistive technology outcome measure captures physical and psychological associated with informal care provision.
Functional Autonomy Measure (Système de mesure de l'autonomie fonctionnelle (SMAF)) | 58 weeks
  A composite from two sub-scales of the SMAF will be used the primary outcome measure for users (self-care and mobility)

SECONDARY OUTCOMES:
Sub-scale scores from the Functional Autonomy Measure (Système de mesure de l'autonomie fonctionnelle (SMAF)) | baseline (Time 0), week 6 (Time 1), week 22 (Time 2) and at week 58 (Time 3)
  Three sub-scales from the Functional Autonomy Measure (Système de mesure de l'autonomie fonctionnelle (SMAF)) (self-care, mobility and instrumental) will be used as secondary outcome measures for assistance users.
Sub-scale scores from the Caregiver Assistive Technology Outcome Measure | baseline (Time 0), week 6 (Time 1), week 22 (Time 2) and at week 58 (Time 3).
  For caregivers, sub-scale scores of frequency of physical and psychological burden from the CATOM will be used.
Euro-QOL 5 | baseline (Time 0), week 6 (Time 1), week 22 (Time 2) and at week 58 (Time 3).
  For caregivers, health-related quality of life. Health related quality of life will be measured using the EuroQol,
Caregiver Burden Inventory | baseline (Time 0), week 6 (Time 1), week 22 (Time 2) and at week 58 (Time 3).
  A composite score from the first three subscales of the Caregiver Burden Inventory will be used as a secondary outcome measure for caregivers.
Reintegration to Normal Living Index (RNLI) | baseline (Time 0), week 6 (Time 1), week 22 (Time 2) and at week 58 (Time 3).
  The RNLI will measure problems with social participation among assistance users.
Self-report of Functional Independence | baseline (Time 0), week 6 (Time 1), week 22 (Time 2) and at week 58 (Time 3).
  Assistance users and caregivers will independently evaluate perceived functional Independence of assistance users.
Qualitative interviews | week 6 and week 58
  A purposive sample of participants will be interviewed immediately after the intervention and at the end of the study to understand better how the intervention was administered by therapists and experienced by assistance users and their caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Louise Demers, PhD, Principal Investigator — Université de Montréal
Locations (3):
- Canada (3):
  - Simon Fraser University- Gerontolgy Research Centre, Vancouver, British Columbia
  - Élisabeth Bruyère Research Centre, Ottawa, Ontario
  - University of Montreal, Montreal, Quebec

REFERENCES:
- [Derived] Ben Mortenson W, Demers L, Fuhrer MJ, Jutai JW, Bilkey J, Plante M, DeRuyter F. Effects of a caregiver-inclusive assistive technology intervention: a randomized controlled trial. BMC Geriatr. 2018 Apr 18;18(1):97. doi: 10.1186/s12877-018-0783-6. PMID 29669536
- [Derived] Demers L, Mortenson WB, Fuhrer MJ, Jutai JW, Plante M, Mah J, DeRuyter F. Effect of a tailored assistive technology intervention on older adults and their family caregiver: a pragmatic study protocol. BMC Geriatr. 2016 May 13;16:103. doi: 10.1186/s12877-016-0269-3. PMID 27177609